CLINICAL TRIAL: NCT02706249
Title: A Randomized, Phase II Study Of Weight-Based Versus Standard Dose Enoxaparin Thromboprophylaxis In High-Risk Hospitalized Cancer Patients
Brief Title: Study Of Weight-Based Versus Standard Dose Enoxaparin Thromboprophylaxis In High-Risk Hospitalized Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeffrey Zwicker, MD, Jeffrey Zwicker, MD, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-547
Record Dates: First submitted 2016-03-03; First posted 2016-03-11 (Estimated); Results first posted 2021-06-10 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Venous Thormboembolism
MeSH Terms: interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Standard Dose Enoxaparin (Active Comparator): Participants will receive Enoxaparin 40 mg subcutaneously once daily. On study Enoxaparin will be administered for up 14 days during hospitalization.
  After the day 14 assessment, treatment arms will be un-blinded in order to appropriately schedule a bilateral lower extremity ultrasound for participants enrolled onto Arm A at day 17.
  Interventions: Drug: Enoxaparin
- B: Weight Adjusted Enoxaparin (Active Comparator): Participants will receive Enoxaparin at 1mg/kg subcutaneously once daily with maximum dose of 100 mg daily. Participants who weigh more than 100kg will be capped at 100mg.
  On study Enoxaparin will be administered for up 14 days during hospitalization.
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin
  Other Names: Lovenox

SUMMARY:
Hospitalized patients with histologically or cytologically confirmed diagnosis of solid tumor malignancy, lymphoma, or multiple myeloma and who are at high risk for a venous thromboembolism will be randomized to standard dose versus intermediate dose enoxaparin.

DETAILED DESCRIPTION:
In a phase II trial, high risk hospitalized cancer patients will be enrolled and randomized to standard dose enoxaparin versus intermediate dose (weight adjusted) enoxaparin thromboprophylaxis. Study subjects will be administered enoxaparin during hospitalization in a double-blinded manner. Following completion of 14 days, the study arms will be unblinded and lower extremity ultrasound performed on the standard dose enoxaparin arm in order to more accurately determine the overall cumulative incidence of thrombosis in this group.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed diagnosis of solid tumor malignancy, lymphoma or multiple myeloma.
* Cancer diagnosis or received treatment (chemotherapy or radiotherapy) for malignancy within the previous 6 months
* One or more Padua-based risk factor:

  * History of previous venous thromboembolic event (excluding superficial vein thrombosis)
  * Reduced mobility (ECOG performance status 3 or 4, see Appendix A)
  * Established hereditary thrombophilia (e.g. Factor V Leiden, G20210 prothrombin mutation, protein C or S deficiency, antithrombin deficiency).
  * Recent surgery within the last 30 days
  * Age ≥ 70 years
  * Congestive heart failure (NYHA class III or IV)
  * Complicated respiratory insufficiency (defined as an increased requirement for supplementary oxygen of at least 2L)
  * Acute myocardial infarction or ischemic stroke
  * Obesity (BMI ≥ 30)
  * Receiving hormonal agents (e.g. tamoxifen, estrogen, testosterone)
  * Acute infection (i.e. requiring antimicrobial therapy)
* Age ≥ 18 years
* Life expectancy of greater than 30 days
* Platelet count ≥ 100,000/mcL
* Creatinine < 1.5 mg/dL or estimated creatinine clearance ≥ 50 mL/min/1.73 m2
* Ability to understand and the willingness to sign a written informed consent document
* Weight between 50kg to 130 kg.

Exclusion Criteria:

* History of allergic reactions attributed to heparin or low molecular weight heparin
* Active bleeding or otherwise considered high risk for hemorrhage (e.g. known acute gastrointestinal ulcer)
* Any history of significant hemorrhage (requiring hospitalization or transfusion) within the last 6 months (excluding hemorrhage during operative procedure).
* History of heparin induced Thrombocytopenia
* Presence of coagulopathy (PT or PTT> 1.2 x upper limit of normal)
* Known diagnosis of disseminated intravascular coagulation
* Currently receiving therapeutic anticoagulant therapy or dual antiplatelet therapy (eg. aspirin and clopidogrel)
* Uncontrolled arterial hypertension (systolic blood pressure > 200mmHg, diastolic >110mmHg)
* Active peptic ulcer disease
* Bacterial Endocardititis
* Received any type of Pharmacologic Thromboprophylaxis (e.g. low molecular weight heparin or heparin) for >48 hours during current hospitalization
* Known brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-04; Primary Completion 2020-12-07 (Actual); Study Completion 2021-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Zwicker, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Cleveland Clinic Foundation, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zwicker JI, Roopkumar J, Puligandla M, Schlechter BL, Sharda AV, Peereboom D, Joyce R, Bockorny B, Neuberg D, Bauer KA, Khorana AA. Dose-adjusted enoxaparin thromboprophylaxis in hospitalized cancer patients: a randomized, double-blinded multicenter phase 2 trial. Blood Adv. 2020 May 26;4(10):2254-2260. doi: 10.1182/bloodadvances.2020001804. PMID 32442298

RESULTS

PARTICIPANT FLOW:
Groups:
- A: Standard Dose Enoxaparin: Participants will receive Enoxaparin 40 mg subcutaneously once daily. On study Enoxaparin will be administered for up 14 days during hospitalization.
  After the day 14 assessment, treatment arms will be un-blinded in order to appropriately schedule a bilateral lower extremity ultrasound for participants enrolled onto Arm A at day 17.
  Enoxaparin
- B: Weight Adjusted Enoxaparin: Participants will receive Enoxaparin at 1mg/kg subcutaneously once daily with maximum dose of 100 mg daily. Participants who weigh more than 100kg will be capped at 100mg.
  On study Enoxaparin will be administered for up 14 days during hospitalization.
  Enoxaparin
Period: Overall Study
Arm/Group | A: Standard Dose Enoxaparin | B: Weight Adjusted Enoxaparin
Started (Patients consented) | 25 | 25
Completed (Evaluated for VTE and safety) | 23 | 24
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Standard Dose Enoxaparin | B: Weight Adjusted Enoxaparin | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants] — Population: Evaluated for VTE and safety
  Participants
    number analyzed (Participants) | 23 | 24 | 47
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 14 | 16 | 30
    >=65 years | 9 | 8 | 17
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Evaluated for VTE and safety
  Participants
    number analyzed (Participants) | 23 | 24 | 47
    Female | 19 | 11 | 30
    Male | 4 | 13 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Evaluated for VTE and safety
  Participants
    number analyzed (Participants) | 23 | 24 | 47
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 2 | 3
    White | 19 | 18 | 37
    More than one race | 1 | 0 | 1
    Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Count of Participants; unit: Participants] — Population: Evaluated for VTE and safety
  Participants
    United States: number analyzed (Participants) | 23 | 24 | 47
    United States | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Venous Thromboembolic Events (VTE) in Standard Dose Enoxaparin Arm at 17 Days
Description: To investigate the numbers of VTE in hospitalized cancer patients receiving standard dose
Time Frame: 17 days only measured in Arm A (Standard dose enoxaparin)
Population: All patients who were randomized to the standard dose of enoxaparin
Measure: Number; unit: participants
Groups:
- A: Standard Dose Enoxaparin: Participants will receive Enoxaparin 40 mg subcutaneously once daily.
Arm/Group | A: Standard Dose Enoxaparin
Number analyzed (Participants) | 23
participants | 2

2. Primary Outcome: Number Participants With Major Hemorrhage
Description: Number of major hemorrhage in weight-adjusted enoxaparin arm and standard-dose enoxaparin arm
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Groups:
- B: Weight Adjusted Enoxaparin: Participants will receive Enoxaparin at 1mg/kg subcutaneously once daily with maximum dose of 100 mg daily
Arm/Group | A: Standard Dose Enoxaparin | B: Weight Adjusted Enoxaparin
Number analyzed (Participants) | 23 | 24
Participants | 1 | 0

3. Secondary Outcome: Number of Symptomatic Venous Thromboembolic Events (VTE)
Description: Comparing number of symptomatic VTE (data collected prior to unblinding) for the standard dose (Arm A) versus intermediate dose enoxaparin (Arm B).
Time Frame: 14 days
Population: The analysis data set is comprised of evaluated patients.
Measure: Count of Participants; unit: Participants
Groups:
- A: Standard Dose Enoxaparin: Participants will receive Enoxaparin 40 mg subcutaneously once daily. .
Arm/Group | A: Standard Dose Enoxaparin | B: Weight Adjusted Enoxaparin
Number analyzed (Participants) | 23 | 24
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events data were collected from the time of the first dose (Day 1) of the study treatment, throughout the study, and until the final study visit (Day 14)
Description: All serious adverse events that occur after the initial dose of study treatment, during treatment, or within 30 days of the last dose of treatment must be reported to the Overall Principal Investigator.
Arm/Group | A: Standard Dose Enoxaparin | B: Weight Adjusted Enoxaparin
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 10/23 | 6/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Standard Dose Enoxaparin (N=23) | B: Weight Adjusted Enoxaparin (N=24)
Skin Infections (Infections and infestations) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Platelets Count Decrease (Investigations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Distal deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pain - extremeties (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Vascular disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Neutrophil Count Decrease (Investigations) | 1 (1) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
GI-Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) — One participant randomly assigned to fixed-dose enoxaparin developed a grade 2 laryngeal bleed occurring several days after completing the trial. the last dose of enoxaparin.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/49/NCT02706249/Prot_SAP_000.pdf